CLINICAL TRIAL: NCT03331289
Title: SGLT2 INHIBITION AND STIMULATION OF ENDOGENOUS GLUCOSE PRODUCTION [EGP]: Can the Glucagon-like Peptide-1 [GLP-1] Receptor Agonist, Exenatide, Prevent the Increase in EGP in Response to Dapagliflozin-induced Increase in Glucosuria
Brief Title: Can Exenatide Prevent Increase in EGP in Response to Dapagliflozin-induced Increase in Glucosuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20170582H; R01DK107680 (NIH)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; dapagliflozin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four groups (20 per group): i) placebo; (ii) exenatide 5 ug subcutaneously; (iii) dapagliflozin (10 mg); and (iv) dapagliflozin 10 mg plus exenatide 5 ug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo (Placebo Comparator): we will examine whether the coadministration of exenatide plus dapagliflozin will prevent the increase in EGP and result in an additive or even synergistic decrease in plasma glucose conc compared to each agent alone.
  Interventions: Drug: Placebo
- Exenatide (Active Comparator): we will examine whether the coadministration of exenatide plus dapagliflozin will prevent the increase in EGP and result in an additive or even synergistic decrease in plasma glucose conc compared to each agent alone.
  Interventions: Drug: Exenatide
- Dapagliflozin (Active Comparator): we will examine whether the coadministration of exenatide plus dapagliflozin will prevent the increase in EGP and result in an additive or even synergistic decrease in plasma glucose conc compared to each agent alone.
  Interventions: Drug: Dapagliflozin
- Exenatide and Dapagliflozin (Active Comparator): we will examine whether the coadministration of exenatide plus dapagliflozin will prevent the increase in EGP and result in an additive or even synergistic decrease in plasma glucose conc compared to each agent alone.
  Interventions: Drug: Exenatide and Dapagliflozin

INTERVENTIONS:
Drug: Placebo — Placebo will be administered to 20 subjects after a 3 hour tracer equilibration period
  Other Names: Placebo drug
  Arms: Placebo
Drug: Exenatide — Exenatide will be administered to 20 subjects after a 3 hour tracer equilibration period
  Other Names: Byetta, Bydureon
  Arms: Exenatide
Drug: Dapagliflozin — Dapagliflozin will be administered to 20 subjects after a 3 hour tracer equilibration period
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Exenatide and Dapagliflozin — Exenatide and Dapagliflozin will be administered to 20 subjects after a 3 hour tracer equilibration period
  Other Names: Byetta plus Dapagliflozin
  Arms: Exenatide and Dapagliflozin

SUMMARY:
Research Design/Plan: After screening, each subject will receive 1 measurements of Endogenous Glucose Production [EGP] with prime-continuous Infusion of 3-3H-glucose. After completing the EGP measurement each subject will receive a Double Tracer Oral Glucose Tolerance Test [OGTT].

Methods: Visit 1: Screening. Medical history will be obtained, physical exam performed, and pregnancy test performed.

Visit 2: Endogenous Glucose Production Measurement: The rate of EGP will be measured with 3-3H-glucose.

Visit 3: Double Tracer OGTT

DETAILED DESCRIPTION:
Eligible subjects will receive a measurement of endogenous glucose production (EGP) with a prime-continuous infusion of 3-3H-glucose. The EGP measurement will be performed in the morning after a 10-12 hour overnight fast and will last 8 hours (from 6 AM to 2 PM). After a 3-hour tracer equilibration period, subjects (20 per group) will receive one of the following medications: (i) placebo; (ii) exenatide 5 ug subcutaneously; (iii) dapagliflozin (10 mg); and (iv) dapagliflozin 10 mg plus exenatide 5 ug. Following the test medication at 9 AM, blood samples will be drawn every 15 minutes for an additional 5 hours and plasma glucose, insulin, C-peptide, glucagon, cortisol, growth hormone, and catecholamine concentrations and glucose specific activity will be measured.

Visit 1: Screening. Medical history & physical exam will be performed. Blood will be drawn for fasting plasma glucose [FPG], routine blood chemistries, complete blood count [CBC], lipid profile, HbA1c, and thyroid function [TSH], Urinalysis, electrocardiogram [EKG], albumin/creatinine ratio and pregnancy test will be performed.

Visit 2: EGP Measurement: The rate of endogenous glucose production will be measured with 3-3H-glucose infusion. [3-3H]-glucose infusion will be started at 6 in the morning [AM] and continued until 2:30 afternoon [PM](5 hours after drug administration). At 6 AM a catheter will be placed into an anticubital vein and a prime (40 uCi x FPG/100)- continuous (0.4 uCi) infusion of [3-3H]- glucose will be started and continued until 2:30 PM. (5 hours after drug administration). Participant's hand will be placed in a box heated to 50-60°C (122-140°F). Baseline blood samples will be obtained at-210, -60, -50, -45, -40, -35, -30, -20, -10, and 0 . After 3.5 hours of tracer equilibration blood samples will be obtained every 10-20 minutes from 9 AM to 2 PM. Plasma glucose, insulin, C-peptide, glucagon, cortisol, growth hormone, and catecholamine concentrations, and [3-3H]-glucose specific activity will be measured. Urine will be collected from 6 to 9 AM and from 9 AM to 2 PM. Urinary volume and glucose concentration will be measured and urinary glucose excretion rate calculated. The study will end at 2:30 PM.

Visit 3: Double Tracer Oral Glucose Tolerance Test [OGTT]: Within the week after the measurement of EGP, all subjects will have a 5-hour OGTT with measurement of plasma glucose, insulin (I), C-peptide (CP), and glucagon concentrations at -180, -6-, -5-, -45, -40, -35, -30, -20, -10, 0 and every 15-30 minutes thereafter to obtain a measure of overall glucose tolerance, insulin secretion (CP0-120/G0-120), insulin sensitivity ([Matsuda Index=MI]), beta cell function, (CP0-120/G0-120 x MI), and suppression of plasma glucagon concentration (64). At 7 AM a catheter will be placed into an antecubital vein and a prime (25 uCi x FPG/100)- continuous (0.25 uCi) infusion of [3-3H]- glucose will be started and continued until 3 PM. Urinary volume and glucose concentration will be measured and urinary glucose excretion rate calculated.

HbA1c will be measured 2x, 1 on the day of the OGTT & 1 on the day of the EGP measurement.

ELIGIBILITY:
Inclusion Criteria:

* Health Status: Type 2 Diabetes Mellitus according to ADA criteria (subjects must be in good general health as determined by physical exam, medical history, blood chemistry-CBC, TSH, T4, EKG and urinalysis)
* BMI: 21-45kg/m
* HbA1C>7.0% and <10.5%
* Medication: Drug naïve and/or on a stable dose of metformin and/or sulfonylurea (more than 3 months)

Exclusion Criteria:

* Health Status: Type 1 Diabetics
* Proliferative diabetic retinopathy
* Plasma Creatinine greater than 1.4mg/dL in females or greater than 1.5mg/dL in males, or 24 hour urine albumin excretion greater than 300mg/dL
* Medication: Subjects taking drugs known to affect glucose metabolism (other than metformin and sulfonylurea)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Health System Texas Diabetic Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared once study closes to enrollment and all data are analyzed and published. Informed consent documentation will be available for sharing.....
Access Criteria: Access will be available through the journal website and on request through the PI.

REFERENCES:
- [Derived] Alatrach M, Agyin C, Solis-Herrera C, Lavryneko O, Adams J, Gastaldelli A, Triplitt C, DeFronzo RA, Cersosimo E. Dapagliflozin Impairs the Suppression of Endogenous Glucose Production in Type 2 Diabetes Following Oral Glucose. Diabetes Care. 2022 Jun 2;45(6):1372-1380. doi: 10.2337/dc21-1798. PMID 35235659

RESULTS

PARTICIPANT FLOW:
Groups:
- Type 2 Diabetes on Dapagliflozin: Patients will be randomized to receive dapagliflozin 10 mg daily, acutely and for 34 months.
- Type 2 Diabetes on Oral Placebo: Randomly selected group of patients with type 2 diabetes who will receive oral placebo for dapagliflozin at the same dosing schedule as dapagliflozin
- Type 2 Diabetes on Exenatide: patients ill be randomized to receive exenatide injections subcutaneously acutely and daily for 4 months.
- Type 2 Diabetes on Exenatide Plus Dapagliflozin: patients will be randomized to receive exenatide injections plus dapagliflozin acutely and for 4 months.
Period: Overall Study
Arm/Group | Type 2 Diabetes on Dapagliflozin | Type 2 Diabetes on Oral Placebo | Type 2 Diabetes on Exenatide | Type 2 Diabetes on Exenatide Plus Dapagliflozin
Started | 30 | 23 | 28 | 26
Completed | 25 | 15 | 25 | 25
Not Completed | 5 | 8 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Exenatide | Dapagliflozin | Exenatide and Dapagliflozin | Total
Number analyzed (Participants) | 15 | 25 | 25 | 25 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (3) | 52 (3) | 51 (2) | 49 (2) | 51 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 17 | 15 | 16 | 58
  Male | 5 | 8 | 10 | 9 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 15 | 14 | 16 | 56
  Not Hispanic or Latino | 2 | 10 | 11 | 9 | 32
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 9 | 8 | 28
  White | 9 | 18 | 16 | 17 | 60
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
ENDOGENOUS GLUCOSE PRODUCTION [EGP] [Mean (Standard Deviation); unit: mg/kg.min] | 2.30 (0.05) | 2.33 (0.13) | 2.27 (0.04) | 2.41 (0.10) | 2.33 (0.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in EGP From Baseline to Post-oral Glucose Load.
Description: The difference in rate of EGP during the last hour of the study (from 240-300 minutes) between drug-treatment and placebo treatment studies represents the effect of drug treatment on EGP, which will be compared among the 3 acute drug treatments (exenatide; dapagliflozin; exenatide plus dapagliflozin this data includes change in EGP above baseline following dapagliflozin alone vs dapagliflozin/exenatide) with ANOVA.
Time Frame: From baseline [-35 to 0min] to the last hour post-glucose load [240-300 minutes]
Population: Type 2 diabetes
Measure: Mean (Standard Error); unit: mg/kg.min
Arm/Group | Placebo | Exenatide | Dapagliflozin | Exenatide and Dapagliflozin
Number analyzed (Participants) | 15 | 25 | 25 | 25
mg/kg.min | -0.03 (0.02) | -0.18 (0.02) | 0.14 (0.03) | -0.08 (0.03)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Adverse events collected during clinical evaluation and laboratory analyses
Arm/Group | Placebo | Exenatide | Dapagliflozin | Exenatide and Dapagliflozin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/15 | 4/25 | 7/25 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=15) | Exenatide (N=25) | Dapagliflozin (N=25) | Exenatide and Dapagliflozin (N=25)
Genital Mycosis (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 4 (4) — Fungal proliferation in the vaginal tract/urethra
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) — nausea and vomiting following subcutaneous administration of exenatide

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT03331289/Prot_SAP_000.pdf